CLINICAL TRIAL: NCT05527275
Title: A Multicenter, Single-arm, Prospective Phase I/II Trial of Mitoxantrone Hydrochloride Liposome Injection Combined With Chidamide in Relapsed or Refractory Peripheral T-cell Lymphoma
Brief Title: A Phase I/II Study of Mitoxantrone Liposome Combined With Chidamide in Relapsed/Refractory Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-140-内科
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Relapsed and Refractory Peripheral T-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection Combined With Chidamide (Experimental)
  Interventions: Drug: Mitoxantrone liposome combine with Chidamide

INTERVENTIONS:
Drug: Mitoxantrone liposome combine with Chidamide — Mitoxantrone Hydrochloride Liposome Injection： Grade 1: 14mg/ m2, D1; Grade 2: 17mg/ m2, D1; Grade 3: 20mg/ m2, D1; Chidamide：20mg twice a week (D1 and D4 or D2 and D5 or D3 and D6) Every 28 days for a cycle, a maximum of 6 cycles of treatment. Mitoxantrone Hydrochloride Liposome Injection RP2D was determined in the phase I trial, and the combination regimen will be used to in the phase II study, with a cycle of every 28 days and a maximum of 6 cycles of treatment.
  Subsequently, maintenance treatment was performed: Chidamide, 20mg twice a week, for 1 year.

SUMMARY:
Peripheral T-cell lymphoma (PTCL) is a highly heterogeneous group of aggressive non-Hodgkin lymphoma (NHL) originating from mature thymus T cells.Mitoxantrone Hydrochloride Liposome Injection can accelerate the entry of mitoxantrone into cells, reduce the efflux of mitoxantrone, ensure the concentration of intracellular drugs, reverse the drug resistance mechanism, and enhance anti-tumor activity.We will explore the dose-limiting toxicity (DLT) of Mitoxantrone Hydrochloride Liposome Injection combined with Chidamide in the treatment of relapsed or refractory peripheral T-cell lymphoma, estimate the maximum tolerated dose (MTD) of the combination, and determine the phase II recommended dose RP2D.In the phase II study, we will evaluate the safety and efficacy of the combination regimen.

DETAILED DESCRIPTION:
This study was a single-arm, open, multicenter phase I/II clinical study. An estimated 87 to 96 patients with relapsed or refractory PTCL will be enrolled. This program is divided into two parts:

The phase I study is expected to enroll 9 to 18 patients with relapsed or refractory PTCL who will be treated with Mitoxantrone Hydrochloride Liposome Injection combined with Chidamide.The phase II study is expected to enroll 78 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients participated voluntarily and signed informed consent；
* PTCL confirmed by histopathology；
* There must be at least one evaluable or measurable lesion that meets Lugano2014 criteria；
* The ECOG score is 0 to 1；
* ANC≥1.5×10*9/L，PLT≥75 × 10*9/L；HB≥80 g/L；TBIL≤1.5ULN；ALT or AST≤2.5 ULN； Scr≤1.5ULN；
* Use contraception during treatment and for one year after the end of treatment.

Exclusion Criteria:

* Patients with central nervous system (CNS) involvement and/or hemophagocytic syndrome；
* The estimated survival time is less than 6 months；
* History of allergy to anthracyclines or liposomes; Previous recipients of mitoxantrone or mitoxantrone liposome;Previous treatment with doxorubicin or other anthracyclines had a cumulative dose of doxorubicin > 360 mg/m2（For other anthracyclines, 1 mg of doxorubicin is equivalent to 2 mg of epirubicin, and the maximum cumulative dose of liposomal doxorubicin is 2460mg/m2）；
* The use of Chidamide is contraindicated;
* Impaired heart function or significant heart disease;
* Hepatitis B, hepatitis C active stage infection;
* Had undergone major surgery within 4 to 6 weeks prior or expected to undergo major surgery during the study;
* severe infection;
* Poorly controlled high blood pressure or diabetes;
* A history of active visceral bleeding within the previous 3 months
* A history of malignancy within five years;
* History of mental illness;
* A history of substance abuse or dependence;
* pregnant or lactating woman;
* The investigators did not consider it appropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
RP2D | 24 months
  Phase II recommended dose
ORR | 24 months
  Objective remission rate

SECONDARY OUTCOMES:
MTD | 24 months
  Maximum tolerated dose
DLT | 24 months
  Dose-limiting toxicity
DOR | 24 months
  Duration of remission time

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology,Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP